CLINICAL TRIAL: NCT01544192
Title: Impact of Oral Versatile Antioxidants on Glaucoma Progression:Comparative Early Results
Brief Title: Impact of Oral Versatile Antioxidants on Glaucoma Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BEAH-Ophthalmol-1
Record Dates: First submitted 2011-10-19; First posted 2012-03-05 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Glaucoma
Keywords: Antioxidant; α-tocopherol; Vitamin E; Gingko Biloba; Glaucoma; Neuroprotection; Retina
MeSH Terms: conditions — Glaucoma | interventions — Ginkgo Extract; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- retinal nerve fiber thickness (Active Comparator)
  Interventions: Drug: Gingko Biloba; Drug: α-tocopherol; Drug: Placebo; Drug: Antioxidant formula
- Mean Deviation (Active Comparator)
  Interventions: Drug: Gingko Biloba; Drug: α-tocopherol; Drug: Placebo; Drug: Antioxidant formula
- Pattern Standard Deviation (Active Comparator)
  Interventions: Drug: Gingko Biloba; Drug: α-tocopherol; Drug: Placebo; Drug: Antioxidant formula
- ganglion cell count (Active Comparator)
  Interventions: Drug: Gingko Biloba; Drug: α-tocopherol; Drug: Placebo; Drug: Antioxidant formula
- c/d ratios (Active Comparator)
  Interventions: Drug: Gingko Biloba; Drug: α-tocopherol; Drug: Placebo; Drug: Antioxidant formula

INTERVENTIONS:
Drug: Gingko Biloba — 2x60 mg Gingko Biloba (Vega Natural, Konya, Turkey)
  Other Names: Gingko Biloba (Vega Natural, Konya, Turkey)
Drug: α-tocopherol — 2x300 mg α-tocopherol
  Other Names: α-tocopherol (Roche Pharma, Istanbul, Turkey)
Drug: Placebo — control group did not receive oral neuroprotective agent
Drug: Antioxidant formula — 2x1 tablet AOF
  Other Names: AOF (Vega Natural, Konya, Turkey)

SUMMARY:
Background: The significance of retinal ganglion cell protection in the glaucoma led the view that, glaucomatous optical neuropathy can also be considered as a pathology of central nervous system. It is known that α-tocopherol and Gingko Biloba have specific neuroprotective and vasoregulatory activities, in addition to antioxidant effects. In this study, the investigators compared early neuroprotective effects of α-tocopherol and GB with each other as well as control and a strong antioxidant formulation in patients with glaucoma.

Methods: In this non-randomized control trial, 120 eyes of 60 patients with glaucoma were enrolled into the study and divided into 4 groups, each consisting of 30 eyes. Unlike the controls, patients in the 3 antioxidant groups received α-tocopherol, Gingko Biloba and a strong antioxidant formula for 3 months. Central vision field and MD, PSD and OCT as well as thickness of retinal nerve fiber layer, ganglion cell counts and c/d ratios were recorded. The data were compared statistically.

DETAILED DESCRIPTION:
A significant difference was observed between MD, PSD, s-RNFL and m-RNFL levels of groups (p<0.05) (Table 3), but when compared with Groups of Vit E and AOF, MD and s-RNFL levels of the Group GB were significantly low and PSD level was significantly high in the same group. m-RNFL level of the Vit E group was significantly higher than m-RNFL levels of GB, AOF and Control groups (p<0.05, p<0.01). In the comparison of Vitamin E with GB, MD values were found significantly higher and PSD values were significantly low (p<0.05). No statistically significant difference was present between I-RNFL levels of groups (p>0.05). While the difference between c/d levels of groups were highly significant (p<0.01) (Table 3), c/d levels of Vit E and GB groups were found significantly lower than c/d levels of AOF and Control groups (p<0.01). c/d level of the Vit E group is significantly lower than c/d levels of AOF and Control groups (p<0.01). No statistically significant difference was found between c/d levels of other groups (p>0.05).

No statistically significant difference was present between s-GCC and i-GCC levels of groups (p>0.05). A high statistically significant difference was found between m-GCC levels of groups (p<0.01). While highly 201 significant and significant difference were present between m-GCC level of the Vit E Group and m-GCC levels of AOF and Control Groups, respectively, (p<0.01, p<0.05), m-GCC level of the Group GB was significantly higher than that of Group AOF (p<0.05). No statistically significant difference was observed between m-GCC levels of other groups (p>0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received follow-up in our glaucoma polyclinics

Exclusion Criteria:

* Known ocular or systemic concomitant disorders
* Previous glaucoma surgeries
* Antioxidant usage

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kaya N Engin, MD,PhD, Study Director — Bagcilar TRH
Locations (1):
- Bakırköy Şadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)